





### INFORMED CONSENT FORM FOR PERMISSION TO PARTICIPATE IN A RESEARCH STUDY

Title: Use of Probiotics to Reduce Infections and Death and Prevent Colonization with Extended-Spectrum beta-lactamase (ESBL) producing bacteria, among newborn infants in Haydom and surrounding area, Tanzania.

Child's Name......

Principal investigator: Dr Joshua G. Gidabayda, Chief Paediatrician

**LOCATION:** Haydom Lutheran Hospital (HLH)

SPONSOR: Haydom Lutheran Hospital

I am....... a clinical research assistant working for this project, and I would like to inform you about the project. You are asked to participate in this research study because you are expecting a child or have just given birth to one. Before you decide you can talk to anyone whom you feel free to discuss about the study. If there is anything you don't understand, please ask me, and I can explain it. If you have any questions later, you may ask me or any employee in this study.

### **INTRODUCTION**

Probiotics are safe live microorganisms that, when administered in adequate amounts, confer a benefit to human beings. Probiotics are currently widely used in newborns and children in developed world. They have proven beneficial effects in reducing incidence of gut inflammation and death of very preterm infants. The main purpose of this study is to evaluate whether use of probiotics among newborn infants can reduce carriage of resistant bacteria and thus reduce severe infections and death caused by these organisms. This study will take place in areas served by the Haydom Lutheran Hospital, which is Mbulu, Hanang and Mkalama district. The study will include a total of 2000 newborns whose parents reside in the study area.

## **PROCEDURES**

If you agree to participate in this study, we will first assess your child's eligibility to participate in the study. You must be aged over 18 years and long-term residents of Hydom and willing to complete study visits schedules over six months follow-up, which also includes hospitalizations required for compliance of this study protocol. Your newborn baby must have a birth weight of ≥2.0 kg. If you have multiple pregnancy, you will not be eligible for the study. If you are willing to let your child participate in the study, we will ask you some questions about yourself during the pregnancy of this child, your age, previous history of illness and treatment. We will also give an identification card for this study, and you will show it to the doctor/nurse who will be attending you during childbirth. The attending doctor/midwives will inform the research assistant of the study about you. After delivery, your newborn baby will be screened for eligibility into the study, if eligible he/she will be enrolled and allocated to the investigational product that will have to be used five drops once daily for four weeks when the bottle is empty. Some participants will receive the actual product under investigation, while others will receive a product called a placebo, that looks the same but does not contain probiotic. Whether your child gets the intervention, or the placebo is by chance. We do not know if the intervention works and therefore you are not necessarily "better off" to get the intervention or the

ENG Version 2.0: Date 19/12/2021

placebo. We will also gather information about your baby and his/her health, and we will do a follow-up of your baby with three visits for six months. The first visit will be after one week, the second at six weeks and the third at six months. We will also take your baby's stool specimen during 2 of the three visits i.e., 6 weeks and 6 months visit. A phone/tablet computer will be used to collect clinical and demographic information of your baby.

#### **SPECIMEN COLLECTION**

One fecal sample will be collected at six weeks and at six months' visits. For storage and research purposes, the fecal sample will be divided into 3 portions by the research assistant collecting the specimen. Some of these specimens will be transported to Norway for further analysis. Laboratory results from these specimens will not be reported back to you because there is no evidence that these infections without symptoms need to be treated. If your child becomes ill and is hospitalized at Haydom Lutheran Hospital because of fever or presents with signs of infection, an additional stool sample will be obtained.

### **POTENTIAL SIDE EFFECTS**

Dietary supplementation containing live enteric bacteria are usually well tolerated and there is no evidence of an increased risk resulting from probiotic use in healthy children. The side effects that may occur are a temporary increase in gas, bloating, and a change in frequency of stools. There is no need to stop the intervention when these minor side effects occur.

#### **ADVANTAGES**

There is no direct benefit for participating in this study. However, this research will increase our knowledge on how much probiotics can reduce carriage/presence of resistant bacteria, infections and death among newborn infants. In addition, the study will provide CRP analysis, and blood culture if the child has fever and malaria test. Laboratory results will be given to the attending clinician responsible for the care of children to assist in patient management.

### **COMPENSATION**

There will be no compensation given for participation in this study, however, even though the study products are not considered to be medicinal drugs, and studies have so far not revealed any serious adverse effects, study participants will be insured, if unforeseen side effects of the probiotics develop.

### **CONFIDENTIALITY**

We will only collect information directly relevant to this study, and all medical doctors and laboratory workers in this study have pledged secrecy. The data will be stored anonymously, meaning that no one can connect the information to you in-person, the study documents will not include your name or any identifier, but a unique number. If you sign this form, you have given us permission to allow the research staff to use and disclose health information about you to conduct this study. The information created about you may be shared with other institutions doing this study, data and safety monitoring boards, accrediting agencies, Government and local agencies (such as Tanzania National Institute for Medical Research (NIMR), Tanzania Medicine and Medical Devices Authority (TMDA)) overseeing this research.

# PARTICIPATION AND RIGHT TO REFUSE OR WITHDRAW FROM THE STUDY

You can decide not to participate in this study, and you can withdraw from participating at any time. Refusal to participate **or withdrawal from** this study will not interfere with the right of your baby to get medical care like any other patient in any hospital. Any information you provide will be kept confidential.

ENG Version 2.0: Date 19/12/2021

# WHO CAN I CONTACT WITH MORE QUESTIONS ABOUT THIS RESEARCH STUDY?

For questions related to the study conduct, feel free to contact: Dr Joshua G. Gidabayda Department of Paediatrics at Haydom Lutheran Hospital, Phone:+255784995669, Email: joggs 2003@yahoo.com, Study Coordinator Dr. Museveni N Justine, Phone Number: +255621043779, Email: museveni.justine@gmail.com, Haydom Lutheran Hospital institution Phone number: +255 (0) 272533194/5. Institution E-mail: post@haydom.co.tz

## WHO CAN I CONTACT WITH QUESTIONS ABOUT MY RIGHTS AS A RESEARCH SUBJECT?

For questions related to your rights as a research participant, contact The National Institute for Medical Research (NIMR); 2448, Ocean Road, P.O.BOX 9653, Dar es salaam, Tanzania, Tel: +255-22-2121400. Email; hq@nimr.or.tz

**CONSENT**: I have read and understand the information on this form. The information on this form was explained to me and I had a chance to ask questions about this research study and my questions have been answered to my satisfaction. I also understand that participating in this study is completely voluntarily and have the right to withdraw at any time. I understand that when I sign my name below, I agree to participate in this research

Signature or thumb print

| Signature Signature or thumb print Signature | Date Date Date |
|---|---|
| Signature or thumb print | Date |
| Signature | Date |
| Signature | Date |
| may place a thumb print on the Participant Signary place a thumb print on the Participant Signary form was presented or ally in my presence unity to ask any questions he/she had about the eely gave their informed consent to participate the identified individual: | gnature to the e study. |
| IMPARTIAL WITNESS (NAME(S)-CAPITAL LETTER PRINT) | DATE |
| 3 | ent form was presented orally in my presence unity to ask any questions he/she had about the rely gave their informed consent to participate the identified individual: IMPARTIAL WITNESS |

ENG Version 2.0: Date 19/12/2021

Name of participant/Pregnant woman

Date